CLINICAL TRIAL: NCT05618223
Title: Dapagliflozin Effect on Rheumatic Mitral Stenosis
Acronym: Dapa-Rhemis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, An Aldia Asrial, An Aldia Asrial, MD, FIHA (Principal investigator), Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dapa-Rhemis
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Rheumatic Heart Disease; Heart Failure; Mitral Stenosis
Keywords: rheumatic heart disease; mitral stenosis; heart failure
MeSH Terms: conditions — Rheumatic Heart Disease; Heart Failure; Mitral Valve Stenosis | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Pre and post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin group (Experimental): Dapagliflozin 10 mg once a day and standard treatment
  Interventions: Drug: Dapagliflozin
- Control group (No Intervention): Standard treatment only.

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg once daily in addition to standard therapy
  Arms: Dapagliflozin group

SUMMARY:
Rheumatic mitral stenosis remains a health problem in developing countries. Progressive fibrosis of the valves and myocardium is the main pathophysiology that plays an important role. Dapagliflozin has various beneficial effects on the heart by reducing fibrosis, reducing inflammation, and improving patient quality of life. However, the role of this therapy is unknown in patients with rheumatic mitral stenosis.

DETAILED DESCRIPTION:
This study is an open-label study on Rheumatic Mitral Stenosis patients, carried out at Sebelas Maret University Hospital Sukoharjo, Panti Rahayu Hospital Purwodadi, and Permata Bunda Hospital Purwodadi. Researchers divided 36 Rheumatic Mitral Stenosis patients sequentially into two groups, the first was the dapagliflozin group which would receive dapagliflozin 10 mg once a day and standard treatment. And the second group will only get standard treatment. Each patient will be examined on PICP, MMP-1, MMP-1/TIMP-1 ratio, TGF-β, Net atrioventricular compliance index, NT-pro BNP, and Kansas City Cardiomyopathy Questionnaire on day 1 and one month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Severe mitral stenosis by echocardiographic examination of the planimetric method with morphology that supports the etiology of rheumatic
* Heart failure in functional class II-III
* Dapagliflozin naive

Exception Criteria:

* Other significant valve diseases
* Pregnant or breastfeeding
* Unstable hemodynamic conditions including cardiogenic shock
* history of mitral valve replacement/repair or mitral balloon valvuloplasty
* history of hypoglycemia
* eGFR below 25 mmHg
* diffuse pulmonary fibrosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvements of Biomolecular Parameters | 4 weeks
  PICP in pg/ml, MMP-1 in pg/ml, MMP-1/TIMP-1 ratio, TGF-β in pg/ml, NT-ProBNP in pg/ml
Improvements of Clinical Parameters | 4 weeks
  Kansas City Cardiomyopathy Questionnaire (KCCQ) scores are scaled 0-100 (the higher score indicates a better condition)
Improvements of Echocardiography Parameters | 4 weeks
  Net atrioventricular compliance in mL/mmHG, mitral valve gradient in mmHg and mPAP in mmHg

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 4 weeks
  All cause cardiac rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: An Aldia Asrial, MD, Principal Investigator — Universitas Sebelas Maret
Locations (1):
- Sebelas Maret University Hospital, Sukoharjo, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banerjee T, Mukherjee S, Ghosh S, Biswas M, Dutta S, Pattari S, Chatterjee S, Bandyopadhyay A. Clinical significance of markers of collagen metabolism in rheumatic mitral valve disease. PLoS One. 2014 Mar 6;9(3):e90527. doi: 10.1371/journal.pone.0090527. eCollection 2014. PMID 24603967
- [Background] Banerjee T, Mukherjee S, Biswas M, Dutta S, Chatterjee S, Ghosh S, Pattari S, Nanda NC, Bandyopadhyay A. Circulating carboxy-terminal propeptide of type I procollagen is increased in rheumatic heart disease. Int J Cardiol. 2012 Apr 5;156(1):117-9. doi: 10.1016/j.ijcard.2012.01.026. Epub 2012 Feb 1. No abstract available. PMID 22305814
- [Background] Lin YW, Chen CY, Shih JY, Cheng BC, Chang CP, Lin MT, Ho CH, Chen ZC, Fisch S, Chang WT. Dapagliflozin Improves Cardiac Hemodynamics and Mitigates Arrhythmogenesis in Mitral Regurgitation-Induced Myocardial Dysfunction. J Am Heart Assoc. 2021 Apr 6;10(7):e019274. doi: 10.1161/JAHA.120.019274. Epub 2021 Mar 20. PMID 33749310
- [Background] Nassif ME, Windsor SL, Tang F, Khariton Y, Husain M, Inzucchi SE, McGuire DK, Pitt B, Scirica BM, Austin B, Drazner MH, Fong MW, Givertz MM, Gordon RA, Jermyn R, Katz SD, Lamba S, Lanfear DE, LaRue SJ, Lindenfeld J, Malone M, Margulies K, Mentz RJ, Mutharasan RK, Pursley M, Umpierrez G, Kosiborod M. Dapagliflozin Effects on Biomarkers, Symptoms, and Functional Status in Patients With Heart Failure With Reduced Ejection Fraction: The DEFINE-HF Trial. Circulation. 2019 Oct 29;140(18):1463-1476. doi: 10.1161/CIRCULATIONAHA.119.042929. Epub 2019 Sep 16. PMID 31524498
- [Background] Ye Y, Bajaj M, Yang HC, Perez-Polo JR, Birnbaum Y. SGLT-2 Inhibition with Dapagliflozin Reduces the Activation of the Nlrp3/ASC Inflammasome and Attenuates the Development of Diabetic Cardiomyopathy in Mice with Type 2 Diabetes. Further Augmentation of the Effects with Saxagliptin, a DPP4 Inhibitor. Cardiovasc Drugs Ther. 2017 Apr;31(2):119-132. doi: 10.1007/s10557-017-6725-2. PMID 28447181
- [Background] Li G, Zhao C, Fang S. SGLT2 promotes cardiac fibrosis following myocardial infarction and is regulated by miR-141. Exp Ther Med. 2021 Jul;22(1):715. doi: 10.3892/etm.2021.10147. Epub 2021 May 3. PMID 34007324